CLINICAL TRIAL: NCT04733352
Title: Using Omics Technology to Explore the Mechanism of Acupuncture Treatment of Different Acupoints of Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Using Omics Technology to Explore the Mechanism of Acupuncture Treatment of Different Acupoints of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Director, department of acupuncture, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH109-REC3-113
Record Dates: First submitted 2020-10-09; First posted 2021-02-02 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acupuncture Therapy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proximal acupoints of knees (Experimental): GB34, SP9, and EX-LE2
  Interventions: Other: acupuncture
- distal acupoints of knees (Experimental): LI11, HT3, and TE10
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — to conduct acupuncture on different acupoints

SUMMARY:
In recent years, commonly used Omics techniques, including genomics, proteomics, metabolomics, have been applied in the studies on the mechanism of acupuncture effect. In the previous study, "Immediate effects of proximal and distal acupoints on the Radial Pressure Pulse-wave in patients with knee osteoarthritis: a randomized controlled trial", significant changes in the spectral-energy of the pulse wave in the proximal-acupoint treatment group and the distal-acupoint treatment group infer pain relief and blood-flow improvement. The scores of the Visual Analog Scale were decreased, and the passive and active range of knee motions were increased. Both of the proximal and distant acupoints could be used for knee osteoarthritis treatment. To advance the previous work by becoming one treatment, this study will explore if there is any Omics difference resulting from the two acupoints, thus examining the mechanism of curative effect of acupuncture. Additionally, Chinese medical emphasizes the relationship between body constitution and diseases and the dynamic change of pulses and meridians during the disease development. These significances are in agreement with Omics features about organism integrity, dynamic, and complexity. The current study will adopt a Chinese medical body constitution survey, the spectral-energy (SE) changes of the pressure wave from the radial artery, and the pulse energy analysis of Ryodoraku to identify the differences in specific genes, protein, and metabolites of various body constitutions, pulses, changes of the pressure wave, aiming to set up the objectification of Chinese medical diagnosis.

DETAILED DESCRIPTION:
Introduction:

In recent years, commonly used Omics techniques, including genomics, proteomics, metabolomics, have been applied in the studies on the mechanism of acupuncture effect. In the previous study, "Immediate effects of proximal and distal acupoints on the Radial Pressure Pulse-wave in patients with knee osteoarthritis: a randomized controlled trial", significant changes in the spectral-energy of the pulse wave in the proximal-acupoint treatment group and the distal-acupoint treatment group infer pain relief and blood-flow improvement. The scores of the Visual Analog Scale were decreased, and the passive and active range of knee motions were increased. Both of the proximal and distant acupoints could be used for knee osteoarthritis treatment. To advance the previous work by becoming one treatment, this study will explore if there is any Omics difference resulting from the two acupoints, thus examining the mechanism of curative effect of acupuncture. Additionally, Chinese medical emphasizes the relationship between body constitution and diseases and the dynamic change of pulses and meridians during the disease development. These significances are in agreement with Omics features about organism integrity, dynamic, and complexity. The current study will adopt a Chinese medical body constitution survey, the spectral-energy (SE) changes of the pressure wave from the radial artery, and the pulse energy analysis of Ryodoraku to identify the differences in specific genes, protein, and metabolites of various body constitutions, pulses, changes of the pressure wave, aiming to set up the objectification of Chinese medical diagnosis.

Method:

The study will recruit 60 participants, which will be recruited when they meet the Clinical Classification Criteria for KOA, that is knee pain and three out of six symptoms can be found in clinical practices, as recommended by the American College of Rheumatology:(a) any gender aged 50 years or above;(b) have less than 30 minutes of morning stiffness; (c) crepitus on active motion; and (d) bony tenderness;(e) bony enlargement; and (f) no palpable warmth. They will be randomly assigned to two groups: the distal-acupoint treatment group (DG) (LI11, HT3 and TE10 and the proximal-acupoint treatment group (PG) (GB34, SP9 and EX-LE2). The study will last for five weeks. Each week has two sessions, as a total of ten sessions. The participants will have blood tests in the following times: before the first acupuncture, after the fifth acupuncture and the tenth acupuncture, three weeks after the end of treatment. The study design is random and single-blind. The participants The primary outcome will come from the assessment: comparing the expressed differences of the genes, proteins, and metabolites of the two acupoints. The secondary outcome will be from the connection among 1) the expressed differences of the specific genes, proteins, 2) the survey of Chinese medical body constitution, 3) the spectral-energy (SE) changes of the pressure wave from the radial artery, and 4) the Ryodoraku pulse energy.

Expected outcome:

The study will use the principle and techniques of Omics to explore the mechanism of the curative effect caused by acupuncture on different acupoints. It is expected to serve as a bridge to connect between contemporary medical and traditional medical.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be recruited when they meet the Clinical Classification Criteria for KOA, that is knee pain and three out of six symptoms can be found in clinical practices, as recommended by the American College of Rheumatology:

* any gender aged 50 years or above;
* have less than 30 minutes of morning stiffness;
* crepitus on active motion;
* bony tenderness;
* bony enlargement;
* no palpable warmth.

Exclusion Criteria:

* Subjects with malignancy, any acute medical condition, poorly controlled diabetes or hypertension, a motor or sensory nerve defect, blood clotting disease, mental illness, dementia, mental retardation or other abnormal person on the organic mind.
* Subjects with intra-articular solid or hyaluronic acid injection in the past 3 months.
* Subjects have undergone knee surgery, knee trauma, congenital knee deformation, severe knee varus or valgus deformation, or endocrine, metabolic, infectious, inflammatory, secondary degenerative knee arthritis caused by problems with rheumatic immune diseases.
* unable to walk.
* Subjects who are hypersensitive to needles.
* Those who are unwilling to cooperate and sign the subject's consent form after explaining and explaining the clinical trial process and purpose.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
the expressed differences of the genes of the two acupuncture groups. | through study completion, an average of 1 year
  The blood samples will be collected 4 times and analyzed which type of gene by quantitative real time-PCR.
the expressed differences of the proteins of the two acupuncture groups. | through study completion, an average of 1 year
  The blood samples will be collected 4 times and analyzed which type of proteins by Micro-Western Array
the expressed differences of the metabolites of the two acupuncture groups. | through study completion, an average of 1 year
  The blood samples will be collected 4 times and analyzed which type of metabolites by LC-MS/MS.

SECONDARY OUTCOMES:
Assessment of Radial Pressure Pulse-wave | There are two sessions each week. The participants will be measured twice in each session. The first time is 10 minutes before the acupuncture treatment; the second time is 10 minutes later after the acupuncture treatment
  Assessment of Radial Pressure Pulse-wave at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph.
Assessment of meridian energy | There are two sessions each week. The participants will be measured twice in each session. The first time is 15 minutes before the acupuncture treatment; the second time is 15 minutes later after the acupuncture treatment
  Assessment of the energy of twelve meridians before and after the intervention using Ryodoraku.
Range of knee motion | before the first session (which is in the first week), after the tenth session (which is in the fifth week), and the three weeks later after the end of the treatment (which is in the eighth week)
  Range of knee motion will be examined by a goniometer.
Visual analog scale (VAS) | before the first session (which is in the first week), after the tenth session (which is in the fifth week), and the three weeks later after the end of the treatment (which is in the eighth week)
  The intensity of pain is measure using VAS for pain. It is incorporated into the questionnaire with a scale of 0 (no pain) to 10 (worst pain possible)
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | before the first session (which is in the first week), after the tenth session (which is in the fifth week), and the three weeks later after the end of the treatment (which is in the eighth week)
  A questionnaire developed to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
The survey of Chinese medical body constitution | 30 min before the first acupuncture treatment
  The scores of the Chinese medical body constitution can tell the difference of the subjects' physical fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D. & Ph.D., Study Director — China Medical University Hospital
Locations (2):
- Taiwan (2):
  - Yiyuantang Chinese Medicine Clinic, Hsinchu
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No